CLINICAL TRIAL: NCT00062673
Title: Duloxetine Versus Placebo in the Treatment of Elderly Patients With Major Depressive Disorder
Brief Title: Study of Duloxetine in Elderly Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6091; F1J-MC-HMBV
Record Dates: First submitted 2003-06-10; First posted 2003-06-12 (Estimated); Last update posted 2007-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Depression; Cognition
MeSH Terms: conditions — Depression | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Duloxetine
Drug: Placebo

SUMMARY:
A study of the safety and efficacy of duloxetine in elderly patients (greater than 65 years old) with major depressive disorder

DETAILED DESCRIPTION:
Duloxetine 60 mg QD and placebo variable-duration, placebo lead-in period 9 weeks in the acute treatment phase

ELIGIBILITY:
Inclusion Criteria:

* You must be able to visit the doctor's office for clinic visits, tests, and procedures.
* You must have been diagnosed with major depression, and have had at least one other episode in the past.

Exclusion Criteria:

* You have a current or previous major psychiatric disorder other than depression, such as bipolar disorder, schizophrenia, or other psychotic disorder.
* You have taken a drug within the last 30 days that has not been approved for use by governmental authorities.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 311
Dates: Start 2003-03; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of duloxetine 60 mg QD & placebo on cognition during acute treatment phase in elderly patients using a composite cognitive score derived from the Verbal Learning & Recall Test (VLRT)
To compare the efficacy of duloxetine 60 mg QD & placebo on cognition during acute treatment phase in elderly patients using a composite cognitive score derived from the Symbol Digit Substitution Test (SDST)
To compare the efficacy of duloxetine 60 mg QD & placebo on cognition during acute treatment phase in elderly patients using a composite cognitive score derived from 2-Digit Cancellation Test (2DCT)
To compare the efficacy of duloxetine 60 mg QD & placebo on cognition during acute treatment phase in elderly patients using a composite cognitive score derived from the Letter-Number Sequencing Test (LNST)

SECONDARY OUTCOMES:
To compare the efficacy of treatment with duloxetine 60 mg QD and placebo on depression as measured by the Geriatric Depression Scale (GDS)
To compare the efficacy of treatment with duloxetine 60 mg QD and placebo on depression as measured by the 17-item Hamilton Depression Rating Scale (HAMD17) total score
To compare the efficacy of treatment with duloxetine 60 mg QD and placebo on depression as measured by response and remission rates
To compare the efficacy of treatment with duloxetine 60 mg QD and placebo on depression as measured by the Clinical Global Impressions of Severity Scale (CGI Severity) and the HAMD17 subscale scores
To compare the efficacy of treatment with duloxetine 60 mg QD and placebo on the painful physical symptoms of depression, as measured by the Visual Analog Scale for pain (VAS)
To compare the safety of duloxetine 60 mg QD and placebo using information on vital signs, electrocardiograms (ECGs), treatment-emergent adverse events, discontinuation-emergent adverse events, discontinuation rates and laboratory analyses
To assess the impact of treatment with duloxetine 60 mg QD and placebo on quality of life as measured by the Short-Form (SF-36) Health Survey

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middleton, Wisconsin, United States

REFERENCES:
- [Derived] Dodd S, Berk M, Kelin K, Zhang Q, Eriksson E, Deberdt W, Craig Nelson J. Application of the Gradient Boosted method in randomised clinical trials: Participant variables that contribute to depression treatment efficacy of duloxetine, SSRIs or placebo. J Affect Disord. 2014 Oct;168:284-93. doi: 10.1016/j.jad.2014.05.014. Epub 2014 Jun 4. PMID 25080392
- [Derived] Oakes TM, Katona C, Liu P, Robinson M, Raskin J, Greist JH. Safety and tolerability of duloxetine in elderly patients with major depressive disorder: a pooled analysis of two placebo-controlled studies. Int Clin Psychopharmacol. 2013 Jan;28(1):1-11. doi: 10.1097/YIC.0b013e32835b09cd. PMID 23138680
- [Derived] Raskin J, Wiltse CG, Dinkel JJ, Walker DJ, Desaiah D, Katona C. Safety and tolerability of duloxetine at 60 mg once daily in elderly patients with major depressive disorder. J Clin Psychopharmacol. 2008 Feb;28(1):32-8. doi: 10.1097/jcp.0b013e318160738e. PMID 18204338
- [Derived] Wise TN, Wiltse CG, Iosifescu DV, Sheridan M, Xu JY, Raskin J. The safety and tolerability of duloxetine in depressed elderly patients with and without medical comorbidity. Int J Clin Pract. 2007 Aug;61(8):1283-93. doi: 10.1111/j.1742-1241.2007.01476.x. Epub 2007 Jun 22. PMID 17590215
- [Derived] Raskin J, Xu JY, Kajdasz DK. Time to response for duloxetine 60 mg once daily versus placebo in elderly patients with major depressive disorder. Int Psychogeriatr. 2008 Apr;20(2):309-27. doi: 10.1017/S1041610207005649. Epub 2007 Jun 22. PMID 17588276
- [Derived] Raskin J, Wiltse CG, Siegal A, Sheikh J, Xu J, Dinkel JJ, Rotz BT, Mohs RC. Efficacy of duloxetine on cognition, depression, and pain in elderly patients with major depressive disorder: an 8-week, double-blind, placebo-controlled trial. Am J Psychiatry. 2007 Jun;164(6):900-9. doi: 10.1176/ajp.2007.164.6.900. PMID 17541049
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com